CLINICAL TRIAL: NCT00054496
Title: Phase II Study Trial Of Tarceva In Patients With Recurrent/Progressive Glioblastoma Multiforme
Brief Title: Erlotinib in Treating Patients With Recurrent or Progressive Glioblastoma Multiforme
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Cleveland Clinic (Other)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000270723; CCF-IRB-5478
Record Dates: First submitted 2003-02-05; First posted 2003-02-06 (Estimated); Last update posted 2014-01-10 (Estimated); Status verified 2006-12

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: adult glioblastoma; recurrent adult brain tumor; adult giant cell glioblastoma; adult gliosarcoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Glioblastoma; Brain Neoplasms; Gliosarcoma | interventions — Erlotinib Hydrochloride

INTERVENTIONS:
Drug: erlotinib hydrochloride

SUMMARY:
RATIONALE: Erlotinib may stop the growth of cancer cells by blocking the enzymes necessary for cancer cell growth.

PURPOSE: Phase II trial to study the effectiveness of erlotinib in treating patients who have recurrent or progressive glioblastoma multiforme.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the response rate of patients with recurrent or progressive glioblastoma multiforme treated with erlotinib.
* Determine the progression-free and overall survival of patients treated with this drug.

OUTLINE: Patients receive oral erlotinib daily. Treatment continues in the absence of disease progression or unacceptable toxicity.

Patients are followed for survival.

PROJECTED ACCRUAL: A total of 73 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed glioblastoma multiforme

  * Radiographic evidence of recurrence or progression

    * Biopsies to confirm tumor recurrence allowed if a sufficent percentage of cases are confirmed to be recurrent tumor
* Previously treated with optimal radiotherapy and at least 1 cytotoxic chemotherapy regimen

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic

* Bilirubin no greater than 2 times normal
* Alkaline phosphatase no greater than 2 times normal
* ALT no greater than 3 times normal

Renal

* BUN no greater than 1.5 times normal OR
* Creatinine no greater than 1.5 times normal

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No medical condition that would interfere with oral administration of erlotinib
* No other medical or psychiatric illness that would preclude study therapy
* No active infection
* No other malignancy within the past 3 years except surgically cured carcinoma in situ of the cervix or nonmelanoma skin cancer

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No concurrent immunotherapy for brain cancer
* No concurrent biologic therapy for brain cancer

Chemotherapy

* See Disease Characteristics
* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas) and recovered
* No concurrent chemotherapy for brain cancer

Endocrine therapy

* Concurrent glucocorticosteroids allowed
* No concurrent hormonal therapy for brain cancer

Radiotherapy

* See Disease Characteristics

Surgery

* Not specified

Other

* No prior epidermal growth factor receptor (EGFR) inhibitor
* No concurrent EGFR inhibitor
* No other concurrent antineoplastic therapy
* No concurrent anti-epileptic agents other than modest- or non-enzyme-inducing drugs such as the following:

  * Gabapentin
  * Lamotrigine
  * Divalproex
  * Felbamate
  * Levetiracetam
  * Tiagabine
  * Topiramate
  * Zonisamide

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Estimated)
Dates: Start 2002-08

PRIMARY OUTCOMES:
Response rate

SECONDARY OUTCOMES:
Progression-free survival
Overall survival
Efficacy of erlotinib in inhibiting epidermal growth factor receptor (EGFR) signaling
Efficacy of tumor EGFR amplification in predicting response to treatment

CONTACTS AND LOCATIONS:
Overall Officials: Michael A. Vogelbaum, MD, PhD, Study Chair — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio, United States